CLINICAL TRIAL: NCT05213936
Title: Scalp Cooling for Chemotherapy-Induced Alopecia in Patients of Color: A Clinical and Mechanistic Study
Brief Title: Scalp Cooling for Chemotherapy-Induced Alopecia in Patients of Color
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Paxman (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-13614
Record Dates: First submitted 2021-12-02; First posted 2022-01-28 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Hair counts using trichoscopy and photographs will be taken at baseline and at the beginning of each chemotherapy cycle, which will be graded by two independent clinicians blinded to the patient group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Scalp cooling with hairstyle (Experimental): Scalp cooling with hairstyle (braids, twists, cornrows) to minimize hair volume and increase scalp cooling cap to scalp contact
  Interventions: Device: Scalp cooling with hairstyle
- Scalp Cooling with conditioner and water emulsion (Experimental): Scalp cooling after coating hair with conditioner and water emulsion to minimize hair volume and increase scalp cooling cap to scalp contact
  Interventions: Device: Scalp cooling with conditioner and water emulsion
- No Scalp Cooling (No Intervention): Control with no scalp cooling

INTERVENTIONS:
Device: Scalp cooling with hairstyle — Hair will be prepared accordingly for the cooling cap fitting based on which approach the patient prefers: braids/cornrows/twists
  Arms: Scalp cooling with hairstyle
Device: Scalp cooling with conditioner and water emulsion — Hair will be prepared accordingly for the fitting based on which approach the patient prefers: or conditioner and water emulsion to coat the hair.
  Arms: Scalp Cooling with conditioner and water emulsion

SUMMARY:
The purpose of this study is to evaluate hairstyling techniques aimed at increasing efficacy of scalp cooling in the prevention of chemotherapy-induced alopecia, determine scalp cooling effect on persistent chemotherapy-induced alopecia, and elucidate molecular mechanisms and predictive biomarkers associated with scalp cooling success in patients with skin of color receiving chemotherapy for breast or non-small cell lung cancer.

This study is being conducted because prior studies have found scalp cooling to be highly effective in preventing hair loss resulting from chemotherapy. However, minority representation was largely limited in completed trials. A recent study found that scalp cooling devices are less efficacious in patients with skin of color, likely because patients with skin of color have hair is predominantly types 3 (curly) and 4 (kinky), which tend to become bulkier when wet and can interfere with scalp cooling cap fitting. The investigators plan to test two techniques aimed at improving scalp cooling efficacy in patients with skin of color through hairstyling methods that minimize hair volume in order to increase cooling cap to scalp contact: 1) cornrows/braids/twists or 2) water/conditioner emulsion on hair. Preliminary data show that breast cancer patients with type 3 or 4 hair receiving taxane chemotherapy and scalp cooling using these techniques to prepare the hair for scalp cooling cap fitting all experienced hair preservation. Additionally, the investigators will also assess persistent chemotherapy-induced alopecia outcomes and incidence by following patients up to 6 months after completing treatment. Finally, specific gene expression changes in taxane-induced chemotherapy-induced alopecia in vitro have been described previously. The investigators will test the hypothesis that scalp cooling reverses such changes in chemotherapy-induced alopecia, assess for biomarkers predictive for scalp cooling success, and investigate persistent chemotherapy-induced alopecia molecular mechanisms using non-invasive transcriptome sequencing on plucked hair follicles.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. Female
3. Hair type 3 (curly) or type 4 (kinky)
4. Diagnosis of breast cancer or non-small cell lung cancer (NSCLC) or gynecologic cancer stage I-IV
5. Patient will be starting >= 4 cycles of taxane-based chemotherapy treatment for curative intent after enrollment

   a. Concurrent HER, cisplatin, cyclophosphamide therapies and doxorubicin therapies allowed
6. Eastern Cooperative Oncology Group (ECOG) 0-2: fully active, restrictive in physically strenuous activity, ambulatory and capable of self-care

Exclusion Criteria:

1. Hair type other than 3 or 4
2. Male
3. Use of hair weave or extensions without plans to remove
4. Concurrent malignancy including hematologic malignancies (i.e. leukemia or lymphoma)
5. Alopecia Common Terminology Criteria for Adverse Events > grade 1 at baseline
6. Past chemotherapy administration if past treatment was <= 10 years ago
7. History of migraines or cluster headaches, anorexia, severe anemia, uncontrolled diabetes, hepatitis, thyroid dysfunction, cold urticaria, cold agglutinin disease, scalp metastases
8. Planned bone marrow ablation chemotherapy or skull irradiation
9. Pregnant patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Severity of chemotherapy-induced alopecia | 6 months after completing treatment, up to approximately 11 months total (from the start to completion of chemotherapy)
  The severity of chemotherapy-induced alopecia as determined by hair counts with trichoscopy with measurements of hair shaft diameter & follicle density and Common Terminology Criteria for Adverse Events (CTCAE Version 5.0) grading
Patient distress during treatment | 6 months after completing treatment, up to approximately 11 months (from the start to completion of chemotherapy)
  Assessed by the Chemotherapy Alopecia Distress Scale and patient self-assessment of hair growth using Common Terminology Criteria for Adverse Events

SECONDARY OUTCOMES:
Severity of persistent chemotherapy-induced alopecia | 26 weeks (starting after chemotherapy completion)
  The severity of chemotherapy-induced alopecia as determined by hair counts with trichoscopy with measurements of hair shaft diameter & follicle density and Common Terminology Criteria for Adverse Events (CTCAE Version 5.0) grading
Patient distress after treatment | 26 weeks (starting after chemotherapy completion)
  Assessed by the Chemotherapy Alopecia Distress Scale and patient self-assessment of hair growth using Common Terminology Criteria for Adverse Events 26 weeks after chemotherapy completion

OTHER OUTCOMES:
Gene expression changes in chemotherapy-induced and persistent chemotherapy-induced alopecia | 26 weeks (starting after chemotherapy completion)
  Using a non-invasive method of plucked hair follicles, the investigators will interrogate patients' hair follicle transcriptome at 26 weeks after chemotherapy completion to clarify persistent chemotherapy-induced alopecia pathogenesis. The investigators will also identify predictive markers for cooling success through transcriptome profiling on hair follicles before and after chemotherapy in intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Beth McLellan, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States